CLINICAL TRIAL: NCT05216718
Title: Prospective Randomized Controlled Study on Mini-flap Bilateral Axillo-breast Approach Robotic Thyroidectomy : Effect on Postoperative Pain and Sensation
Brief Title: Mini-flap BABA (Bilateral Axillo-breast Approach) Robotic Thyroidectomy is Safe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Dongsik Bae, Associate Professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-10-014-001
Record Dates: First submitted 2021-12-30; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Thyroid Nodule
Keywords: Mini-flap; Bilateral axillo-breast approach; Da vinci; Robot-assisted thyroid surgery
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional flap (Experimental): BABA robotic-thyroidectomy that using conventional flap
  Interventions: Procedure: Conventional flap
- Mini-flap (Active Comparator): BABA robotic-thyroidectomy that using Mini-flap
  Interventions: Procedure: Mini-flap

INTERVENTIONS:
Procedure: Mini-flap — Mini-flap BABA robotic-thyroidectomy creates flaps up to the cricoid cartilage
  Arms: Mini-flap
Procedure: Conventional flap — Conventional flap BABA robotic-thyroidectomy creates flaps up to the thyroid cartilage
  Arms: Conventional flap

SUMMARY:
In this study, a randomized controlled study was conducted between two groups of 40 recipients of conventional flap during BABA robotic-thyroidectomy and 40 recipients of Mini-flap method during BABA robotic-thyroidectomy. In this study, we tried to determine whether the use of Mini-flap can reduce sensory loss and pain after BABA robotic-thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* subjects who will have thyroid surgery
* subjects who has no evidence of lymph node metastasis on palpation and imaging (cN0)
* subjects who has thyroid nodule under 4cm (<cT2)
* subjects who has no distant metastasis (M0)

Exclusion Criteria:

* subjects who has clinical evidence of lymph node metastasis (cN1a or cN1b)
* subjects who has both thyroid nodule
* subjects who underwent any radiotherapy on neck
* subjects who has primary hyperparathyroidism
* subjects who underwent head and neck surgery
* subjects who disagree to do this trial

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-24 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain, as measured by the Visual Analog Score(VAS) | 2, 24, 48, 72 hours after surgery
  Visual Analog Score for pain, range from 0 to 10, Higher the values represents more pains
change from baseline in pain, as measured by the number of analgesics uses | 2, 24, 48, 72 hours after surgery
  number of analgesics(additional ketorolac uses)
change from baseline in Sensory change, as measured by the monofilaments | 1 day before surgery, 1, 3 months after surgery
  Six monofilaments were used to measure the pressure threshold of the 2 chest zones and 2 neck zones

SECONDARY OUTCOMES:
Incidence of vocal cord palsy | before surgery, 1 day after surgery, 2, 6 weeks after surgery, 6 month, 1year after surgery
  Check vocal cord palsy that means injury of the recurrent laryngeal nerve with a direct laryngoscope
change from baseline in Hypoparathyroidism, as measured by parathyroid hormone level | before surgery, 1 day after surgery, 2, 6 weeks after surgery, 6 month, 1year after surgery
  check PTH (parathyroid hormone) level

CONTACTS AND LOCATIONS:
Locations (1):
- Dong sik Bae, Busan, South Korea